CLINICAL TRIAL: NCT03355495
Title: A Randomized Controlled Trial Comparing Right vs Left Lateral Decubitus Positioning on Outcomes in Colonoscopy
Brief Title: R vs L Lateral Decubitus Positioning in Colonoscopy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Memorial University of Newfoundland (Other)
Collaborators: Eastern Health (Other)
Responsible Party: Principal Investigator, Alison Greene, Principal Investigator, Memorial University of Newfoundland
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 2017242
Record Dates: First submitted 2017-11-20; First posted 2017-11-28 (Actual); Last update posted 2022-04-05 (Actual); Status verified 2022-04

CONDITIONS: Colonic Adenoma; Colonic Cancer
Keywords: Colonoscopy; Cecal Intubation Rate
MeSH Terms: conditions — Colonic Neoplasms | interventions — Endoscopy

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Left Lateral Decubitus Position (No Intervention): Gold standard positioning for colonoscopy
- Right Lateral Decubitus Position (Active Comparator): Comparing positioning in Right Lateral Decubitus (intervention) for visualization in colonoscopy to the gold standard of Left Lateral Decubitus.
  Interventions: Procedure: Colonoscopy - Position Change

INTERVENTIONS:
Procedure: Colonoscopy - Position Change — Colonoscopy is the gold standard for detecting precancerous lesions. We are proposing that changing positions will provide better visualization for detecting such lesions. We will test our intervention of patients positioned in the Right Lateral Decubitus Position to the gold standard of Left Lateral Decubitus Positioning, hypothesizing better visualization in the right lateral decubitus position.
  Other Names: Endoscopy
  Arms: Right Lateral Decubitus Position

SUMMARY:
Colonoscopy continues to be the gold standard in detecting precancerous lesions in the colon. It relies on adequate visualization of the bowel wall to see and remove such lesions. Visualization is improved with luminal distention, and a multitude of studies have been done to determine ways to increase this luminal distention. The investigators theorize that positioning in the Right Lateral Decubitus rather than the Left Lateral Decubitus may be a cost free method to increase luminal distention and, hence, improve visualization in colonoscopy. In the Right Lateral Decubitus position, the sigmoid colon and cecum - both parts of the bowel that are not fixed - air used during colonoscopy will rise in a dependent fashion, increasing luminal distention. In the left lateral decubitus position, the bowel collapses, creating an often difficult area to maneuver and visualize. The investigators would like to compare both positions to determine if it affects outcomes in colonoscopy. In particular, cecal intubation rates and adenoma detection rates.

DETAILED DESCRIPTION:
Colonoscopy is considered the gold standard for detecting precancerous lesions in the bowel - providing both diagnostic and therapeutic value. Colonoscopy is, ultimately, operator dependent and relies on adequate visualization of these lesions. A multitude of studies have been done to determine the best way to achieve luminal distention that provides the best visualization to detect and remove adenomas. Recent literature has studied the effect of position changes in colonoscopy. Position changes have been theorized to increase luminal distention in the bowel - improving visualization and maneuverability through the colon. Both air and water are used during colonoscopy, with air rising in a dependent fashion in the colon to the highest point. The standard position to perform colonoscopy is left lateral decubitus. In this position, parts of the bowel collapse as air rises into other parts of the bowel. This includes the sigmoid colon and the cecum, both of which are not fixed and can therefore collapse becoming technically challenging to maneuver around. In the right lateral decubitus position, the air rises into these unfixed areas of bowel and are easier to maneuver. A trial by Vergis et al found that right lateral decubitus resulted in quicker examination times and more comfort in their cohort of patients as opposed to the left lateral decubitus position. The investigators note, however, that the population in which this study took place are not comparable to the patients in Newfoundland and in Canada. The investigators also note a study by Ou et al that found position changes had no effect in adenoma detection. Furthermore, a study by Ball et al found conflicting results with position change increased adenoma detection in the right but not the left side of the colon. Conflicting results between all these trials and the populations used have lead to us question if position changes, a cost free and technically easy intervention, can increase visualization in colonoscopy. The investigators propose a randomized controlled trial that compares positioning patients in the right lateral decubitus or left lateral decubitus to aid in luminal distention and visualization, decreasing cecal intubation time and ultimately increasing adenoma detection rate in colonoscopy.

In this trial, participation in the study will be offered when patients present for their scheduled colonoscopy. The patients will be consented at this time for both the colonoscopy procedure and participation in the trial. Patients who consent to take part will then be randomly assigned to either the right or left lateral decubitus starting position. The colonoscopy will then be done in the usual manner with appropriate sedation. Timing throughout the colonoscopy, the number of polyps found and quality of the visualization will then be recorded during the procedure. Patients will then be debriefed regarding their colonoscopy following the procedure in recovery.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years of age or older presenting for their scheduled colonoscopy

Exclusion Criteria:

* Previous bowel resection
* Unable to stay in either the right or left lateral decubitus position, due to pre-existing musculoskeletal problems, previous hip surgery, etc.
* Refusal to participate
* Inability to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 172 (Estimated)
Dates: Start 2019-03-01 (Actual); Primary Completion 2023-06-30 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
Decrease in Cecal Intubation Time | 3 months
  The time it takes for a colonoscopist to start a colonoscopy and reach the cecum (endpoint or target area)

SECONDARY OUTCOMES:
Increase in Cecal Intubation Rate | 3 months
  An important indicator in colonoscopy quality, the percentage of times a colonoscopist can reach the cecum during colonoscopy.
Increase in Adenoma Detection Rate | 3 months
  The number of adenomas visualized during withdrawal of a colonoscope

CONTACTS AND LOCATIONS:
Overall Officials: Alison M Greene, Medicine, Principal Investigator — Memorial University of Newfoundland
Locations (1):
- Health Sciences Centre, St. John's, Newfoundland and Labrador, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Vergis N, McGrath AK, Stoddart CH, Hoare JM. Right Or Left in COLonoscopy (ROLCOL)? A Randomized Controlled Trial of Right- versus Left-Sided Starting Position in Colonoscopy. Am J Gastroenterol. 2015 Nov;110(11):1576-81. doi: 10.1038/ajg.2015.298. Epub 2015 Sep 29. PMID 26416195
- [Result] Ou G, Kim E, Lakzadeh P, Tong J, Enns R, Ramji A, Whittaker S, Ko HH, Bressler B, Halparin L, Lam E, Amar J, Telford J. A randomized controlled trial assessing the effect of prescribed patient position changes during colonoscope withdrawal on adenoma detection. Gastrointest Endosc. 2014 Aug;80(2):277-83. doi: 10.1016/j.gie.2014.01.032. Epub 2014 Mar 12. PMID 24629419
- [Result] Ball AJ, Johal SS, Riley SA. Position change during colonoscope withdrawal increases polyp and adenoma detection in the right but not in the left side of the colon: results of a randomized controlled trial. Gastrointest Endosc. 2015 Sep;82(3):488-94. doi: 10.1016/j.gie.2015.01.035. Epub 2015 Apr 22. PMID 25910661